CLINICAL TRIAL: NCT04453930
Title: A Single-arm，Open Lable Study of Sequential Therapy of Camrelizumab Combined With Chemotherapy（Irinotecan Plus Platinum）and With Apatinib in Participants With Untreated Advanced Small Cell Lung Cancer（SCLC）
Brief Title: A Study of Sequential Therapy of Camrelizumab Combined With Chemotherapy（Irinotecan Plus Platinum）and With Apatinib in Participants With Untreated Advanced Small Cell Lung Cancer（SCLC）
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Li Zhang, professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-2195
Record Dates: First submitted 2020-06-22; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — camrelizumab; Platinum; Irinotecan; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Irinotecan+Platinum→Camrelizumab+apatinib (Experimental): Participants received intravenous infusions of Camrelizumab 200 mg in combination with carboplatin to achieve an initial target area under the concentration-time curve (AUC) of 5 milligrams per milliliter per minute (mg/mL/min) or Cisplatin 30 milligrams per square meter (mg/m^2) followed by Irinotecan 65 mg/m^2 on Day 1 of every 21-day cycle during the induction phase (Cycles 1-4/5/6). On Days 8 of every 21-day cycle during the induction phase (Cycles 1-4/5/6), Cisplatin 30 mg/m^2 and Irinotecan 65 mg/m^2 was administered. Thereafter, participants received maintenance (Cycle onward) Camrelizumab 200 mg on Day 1 of every 21-day cycle with Apatinib 250mg until persistent radiographic PD, symptomatic deterioration, intolerable toxicity, withdrawal of consent, death, or study termination by the Sponsor.
  Interventions: Drug: Camrelizumab，an engineered anti-PD-1 antibody; Drug: Platinum; Drug: Irinotecan; Drug: Apatinib

INTERVENTIONS:
Drug: Camrelizumab，an engineered anti-PD-1 antibody — Camrelizumab intravenous infusion was administered at a dose of 200 mg on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4/5/6) and maintenance phase (Cycle onward).
  Other Names: SHR-1210
Drug: Platinum — Carboplatin： Carboplatin intravenous infusion to achieve an initial target AUC of 5 mg/mL/min was administered on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4/5/6).
  Cisplatin： Cisplatin intravenous infusion was administered at a dose of 30 milligrams per square meter (mg/m^2) on Day 1，8 of every 21-day cycle during the induction phase (Cycles 1-4/5/6).
Drug: Irinotecan — Irinotecan intravenous infusion was administered at a dose of 65 milligrams per square meter (mg/m^2) on Day 1，8 of every 21-day cycle during the induction phase (Cycles 1-4/5/6).
Drug: Apatinib — Apatinib was administered at a dose of 250 mg during the maintenance phase.

SUMMARY:
This single arm, open label, single center, prospective study was designed to evaluate the safety and efficacy of Sequential Therapy of Camrelizumab (humanized monoclonal antibody against Programmed death 1 [PD-1] ) in combination with Chemotherapy（Irinotecan plus Platinum）and with Apatinib (selective Vascular Endothelial Growth Factor Receptor 2(VEGFR-2) tyrosine kinase inhibitor [TKI]) in chemotherapy-naive participants with SCLC. Participants will receive Camrelizumab + Irinotecan + Platinum on 21-day cycles for 4-6 cycles in the induction phase followed by maintenance with Camrelizumab + Apatinib until progressive disease (PD) as assessed by the investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). Treatment can be continued until persistent radiographic PD or symptomatic deterioration.

ELIGIBILITY:
Inclusion Criteria

1. Extensive small cell lung cancer diagnosed by pathology or cytology.
2. Patients with extensive stage small cell lung cancer who have not previously been treated for tumors (including radiotherapy, chemotherapy, use of similar VEGFR inhibitors and immune checkpoint inhibitors).
3. The disease progress of the patients with limited SCLC who had received chemotherapy/radiotherapy before, and no further treatment more than 6 months after the last chemotherapy/radiotherapy.
4. Expected survival≥3months.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Subjects enrolled must have measurable lesion(s) according to the RECIST 1.1 standard (the CT scan length of the tumor lesion > 10 mm)
7. The main organ function is normal. All baseline laboratory requirements will be assessed and should be obtained within -14 days of randomization. Screening laboratory values must meet the following criteria. a .Hemoglobin ≥ 9.0 g/dL (90 g/L) b .Absolute neutrophil count ≥ 1.5 x 109/L c .Platelets ≥ 100 x 109/L d .Total bilirubin (TBIL) ≤ 1 x upper limit of normal (ULN) e .Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 x upper limit of normal(ULN); alkaline phosphatase ≤ 5 x ULN f .Serum creatinine ≤ 1.5 x ULN or creatinine clearance > 45 mL/minute (using Cockcroft/Gault formula)
8. Emale participants of childbearing potential must have a negative serum pregnancy test within -7 days of randomization and must be willing to use very efficient barrier methods of contraception or a barrier method plus a hormonal method starting with the screening visit through 60 days (about 5 drug half-life + menstrual cycle) after the last dose of SHR-1210. Male participants with a female partner(s) of child-bearing potential must be willing to use very efficient barriermethods of contraception from screening through 120 days (about 5 drug half-life + sperm depletion cycle) after the last dose of SHR-1210.
9. Subjects should be voluntarily participate in clinical studies and informed consent should be signed.

Exclusion Criteria:

1.Imaging (CT or MRI) showed the presence of a central tumor that invades the local large vessels. Or there are obvious pulmonary cavitation or necrotizing tumors. 2. Patients with brain metastasis or meningeal metastasis.

3.Subjects used immunosuppressive drugs excluding nasal spray and inhaled corticosteroids or systemic steroids at physiological doses(prednisolone≤10 mg/day or other corticosteroids of the same pharmacophysiological dose) within 14 days before the first dose.

4.Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite with the optimal medical treatment.

5.Subjects with grade II or above myocardial ischemia or myocardial infarction and poorly controlled arrhythmias (QTc interval > 450 ms for males and QTc interval > 470 ms for females). Subjects with grade III-IV cardiac insufficiency or with left ventricular ejection fraction (LVEF) less than 50% had myocardial infarction within 6 months before admission according to NYHA criteria.

6.Accompanied by uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.

7.Participants who had any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis , Hyperthyroidism, decreased thyroid function).

8.Subjects with childhood asthma has completely resolved, adults can be included without any intervention; subjects with bronchodilators for medical intervention can not be included .

9.Participants who had abnormal blood coagulation (INR>1.5 or PT> ULN+4s, and or APTT > 1.5 ULN), bleeding tendency or receiving thrombolytic or anticoagulation；Note: under the premise that the international standardized ratio of prothrombin time (INR) is ≤ 1.5, the use of low-dose heparin (60,000-12,000u per day for adults) or low-dose aspirin (≤ 100mg per day) is allowed for preventive purposes.

10.Urine routine indicates urinary protein ≥ ++, or confirms that 24-hour urine protein is ≥1.0 g.

11.Patients with non-healing wound, non-healing ulcer, or non-healing bone fracture; 12.The patient has severe infection within 4 weeks before first administration（such as the need for intravenous antibiotics, antifungals or antivirals) and unexplained fever within 7 days before administration, ≥38.5 °.

13.There was significant coughing blood and significant clinically significant bleeding symptoms or a clear tendency to hemorrhage in the first 2 months before enrollment (such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ++ and above at baseline, or suffering from vasculitis, etc.).

14.Serious Arterial / venous thrombosis events, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism, within 12 months before enrollment.

15.Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection. (HBV: HBsAg positive and HBV DNA ≥ 500 IU/mL ; HVC: HCV RNA positive and abnormal liver function). And subjects with active tuberculosis.

16.Patients with a clear history of allergies may be potentially allergic to or intolerant to biological agents such as irinotecan, cisplatin, apatinib, and carillizumab; 17.There are obvious factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction. Or sinus or perforation of empty organs within 6 months.

18.Any known mental illness or substance abuse that may have an impact on compliance with the test requirements.

19.There are other factors lead to patients can not participate in this clinical study by the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) as assessed by RECIST 1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  PFS is defined as the time from date of enrollment to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurs first per RECIST 1.1.
Duration of Overall Survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  OS is defined as the time from date of enrollment to date of death from any cause.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) as assessed by RECIST 1.1 | through study completion, an average of 2 year.
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or stable disease per RECIST 1.1.
Objective Response Rate (ORR) as assessed by RECIST 1.1 | through study completion, an average of 2 year.
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response(CR) or a Partial Response(PR) per RECIST 1.1.
Duration of Response (DOR) as Assessed by the Investigator Using RECIST v1.1 | through study completion, an average of 2 year.
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or stable disease per RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No